CLINICAL TRIAL: NCT01233804
Title: Opting In vs Opting Out: Impact on Influenza Vaccination in Pregnant Women
Brief Title: Opting In vs Opting Out
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Gilstrap, Larry C, M.D. (Individual)
Responsible Party: Principal Investigator, Susan Wootton, Assitant Professor - Ctr For Clnc Rsrch & Evidnc MD, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-10-0557
Record Dates: First submitted 2010-10-27; First posted 2010-11-03 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Influenza Vaccination
Keywords: influenza vaccination rates
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opting in (No Intervention): Currently, pregnant women have to sign a consent stating that they want the influenza vaccine (at the clinics where the study is being conducted). Therefore, this group is the same as usual care. However, women will then be asked if they would like to take part in parts 2 and 3 of the study.
- Opting Out (Experimental): Women will sign a consent form only if they do not want to receive the flu vaccine.
  Interventions: Other: Opting Out

INTERVENTIONS:
Other: Opting Out — Usual care is for pregnant women to sign a consent to get the influenza vaccine. The intervention is to offer a group of women the option to sign only when they refuse the influenza vaccine.
  Arms: Opting Out

SUMMARY:
The purpose of this study is to compare methods for consenting (opting in vs opting out) on influenza vaccine uptake rate in pregnant women. This study is designed to learn about the impact of influenza vaccination in pregnant women. This study will help gather knowledge about influenza vaccine side effects (if given) and whether the vaccine reduces the number of respiratory infection in mothers and their infants.

DETAILED DESCRIPTION:
Pregnant women who present for routine prenatal care when influenza vaccine is available would be eligible. Enrolled women would be randomized to either the Opting in (obtaining written consent to administer the vaccine) or Opting out (signing only to refuse the vaccine) study group (Part 1). Vaccine uptake rate and reason for refusal will be captured for enrollees. At the end of this clinic visit, enrollees will be asked if they are interested in participating in Part 2 and 3 of the study. If yes, consent will be obtained. Part 2 of the study, a random sample of 50 women will be called 2 days after enrollment to determine 1) vaccine side effects 2) recall of information provided in consent and 3) to confirm next followup visit with Obstetrician. During Part 3, at 6 weeks post EDD (estimated due date), data about episodes of respiratory illness in the mothers and their infants occuring between the time when influenza vaccine was offered (Part 1) and 6 weeks post-EDD will be abstracted using a standard form. Data will be collected retrospectively by research nurses.

ELIGIBILITY:
Inclusion Criteria:

* pregnant female age >17 years
* presenting for routine PNC at UT Houston or UT Galveston
* pregnant during influenza season
* pregnant when influenza vaccine available

Exclusion Criteria:

* influenza vaccine contraindication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Vaccination rates | time 0 of part one study visit
  Vaccination rates will be analyzed for the two groups (opting in vs opting out) to determine group vaccination rate.

CONTACTS AND LOCATIONS:
Overall Officials: Susan H Wootton, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - University of Texas Medical Branch, Women's Clinics, Galveston, Texas
  - University of Texas Health Science Center at Houston, Professional Building, Houston, Texas